CLINICAL TRIAL: NCT07013825
Title: Prediction of Emergency Department Admission Volume
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0029.1_URGENCES
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Retrospective cohort. Schedule emergency service overload periods on different terms, by hour or time slot over several days.

ELIGIBILITY:
Minor patients Refusal of inclusion in a study explicitly stated in the medical record Objection to the use of data or refusal to participate No consultation at the emergency department in the year prior to the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study participants will be selected from a population of patients who meet specific inclusion and exclusion criteria. Specifically, the population will consist of individuals who:
  Are adult patients (i.e., not minors),
  Have not refused to be included in the study, as indicated in their medical records,
  Have not objected to the use of their medical data or explicitly refused to participate,
  Have had at least one consultation at the emergency department in the year prior to the study period.
  Thus, the study population will include adult patients with documented emergency department visits in the past year, who have not opted out of data use and have no recorded refusal to participate.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Rate of admissions to emergency rooms | 01/01/2022 - 31/12/2022

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France